CLINICAL TRIAL: NCT02615938
Title: Hydroxychloroquine in Pediatric ILD: START Randomized Controlled in Parallel-group, Then Switch Placebo to Active Drug, and STOP Randomized Controlled in Parallel-Group to Evaluate the Efficacy and Safety of Hydroxychloroquine (HCQ)
Brief Title: Hydroxychloroquine (HCQ) in Pediatric Interstitial Lung Disease (ILD)
Acronym: HCQ-chILD-EU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of ressources after inspection and appropriate correcting actions to be taken
Sponsor: Matthias Griese (Other)
Responsible Party: Sponsor-Investigator, Matthias Griese, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudratCT:2013-003714-40
Record Dates: First submitted 2015-11-08; First posted 2015-11-26 (Estimated); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Interstitial Lung Disease; Diffuse Parenchymal Lung Disease; Children´s Interstitial Lung Disease
Keywords: Childhood ILD; Fibrosing lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Goal of the study was to include all chILD patients who are planned to be, or are actively being, treated with HCQ. The character of this study is explorative. It was designed to closely accommodate the current clinical care situation.The study was an explorative, prospective, randomized, doubleblind, placebo-controlled investigation of HCQ in chILD and was one of the first investigator-initiated trials in this condition. The study contained two different study blocks, a START and a STOP block, which could be initiated in any sequence. Each patient can participate in each block only once. In the START block, subjects were randomized to parallel groups for 4 weeks treatment, then the placebo group switched to the active drug. In the STOP block, subjects taking HCQ were randomized into parallel groups (placebo or HCQ).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-bitter taste, same color and form capsule. Verum-same color, form capsule as placebo
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Start HCQ block Verum (Experimental): 4 weeks of Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., once daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg.
  Then 4 weeks Hydroxychloroquine Sulfate (HCQ, Quensyl). First week loading dose 10 mg/kg bw/d, p.o., once daily in the evening, followed by 6.5 mg/kg bw/d for 3 weeks.
  Interventions: Drug: Hydroxychloroquine sulfate
- Start HCQ block Placebo (Placebo Comparator): 4 weeks of Placebo in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg.
  Then 4 weeks Hydroxychloroquine Sulfate (HCQ, Quensyl). First week loading dose 10 mg/kg bw/d, p.o., once daily in the evening, followed by 6.5 mg/kg bw/d for 3 weeks.
  Interventions: Other: Placebo
- Stop HCQ block Verum (Experimental): Individual dose of Hydroxychloroquine Sulfate (HCQ, Quensyl) 6-10 mg/kg bw/d, p.o., once daily in the evening; the maximum daily dose is 400 mg. The dose on which the patient was included into the trial was continued for 3 months. Then the medication was stopped and the patient followed for additional 3 months.
  Interventions: Drug: Hydroxychloroquine sulfate
- Stop HCQ block Placebo (Placebo Comparator): Individual dose of Placebo 6-10 mg/kg bw/d, p.o., once daily in the evening; the maximum daily dose is 400 mg. The dose on which the patient was included into the trial was continued for 3 months. Then the medication was stopped and the patient wo received HCQ will be followed up for additional 3 months with no medication.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine sulfate — Apply drug to modify lysosomal pH
  Other Names: Quensyl
  Arms: Start HCQ block Verum; Stop HCQ block Verum
Other: Placebo — Apply Placebo not to modify lysosomal pH
  Other Names: no other name
  Arms: Start HCQ block Placebo; Stop HCQ block Placebo

SUMMARY:
This is an exploratory Phase 2, randomized, double-blind, placebo-controlled, parallel-group, multinational study investigating the initiation or withdrawal of hydroxychloroquine in subjects with chILD.

DETAILED DESCRIPTION:
This study is an explorative, prospective, randomized, double-blind, placebo controlled investigation of hydroxychloroquine (HCQ) in pediatric ILD. The treatments are organized in START and STOP blocks, which can be initiated in sequence, as needed by the subjects. Each patient can participate in each block only once. In the START block subjects are randomized to parallel-groups, then the placebo group is switched to active drug. In the STOP block, subjects on HCQ are randomized into parallel-groups treated with placebo or HCQ to investigate the withdrawal of HCQ for assessment of its efficacy.

ELIGIBILITY:
Inclusion criteria:

1. Patients should be clinically stable during baseline (between Visit 1 and 2) for inclusion into the study

   1. To determine this, attending physicians can use SpO2 in room air for patients on room air or on O2-supplement; the absolute difference on SpO2 is expected not to be ≥ 5% between Visit 1 and 2. For patients on respiratory support, the summary key parameters should not change ≥ 20% between Visit 1 and 2 and
   2. No major changes in other medications between Visit 1 and 2
2. Mature newborn ≥ 37 weeks of gestation, age ≥ 3 wks and <2y or Infants and children (≥2y and < 18y) or Adults (≥18 and ≤30y) or Previously preterm (≤ 37 weeks of gestation) babies or children and adults of all ages if chILD genetically diagnosed (see inclusion criterion 3.)
3. Diagnosis of chronic (≥ 3 wks of duration) diffuse parenchymal lung disease (DPLD = chILD), defined in at least one of the following ways:

   1. chILD genetically diagnosed surfactant dysfunction disorders including patients with mutations in SFTPC, SFTPB, ABCA3, TTF1 (Nkx2-1), further extremely rare entities with specific mutations, for example in TBX4, NPC2, NPC1, NPB, COPA, LRBA and other genes. In this case, also previously preterm (≤ 37 weeks of gestation) babies or children and adults of all ages can be included into the study.
   2. chILD histologically diagnosed

      * Chronic pneumonitis of infancy (CPI)
      * Desquamative interstitial pneumonia (DIP)
      * Lipoid pneumonitis / Cholesterol pneumonia
      * Nonspecific interstitial pneumonia (NSIP)
      * PAP after the exclusion of mutations in GMCSF-Ra/b and GMCSF autoantibodies*
      * Usual interstitial pneumonia (UIP)
      * Follicular bronchitis/bronchiolitis/Lymphocytic interstitial pneumonia (LIP)
      * Storage disease with primary pulmonary involvement (e.g. Niemann Pick)
      * Hermansky-Pudlak Syndrome
      * Idiopathic pulmonary haemorrhage (haemosiderosis)*
      * Other histology diagnosing chILD, in particular combination of the above pattern, but not exclusively
4. Start block: no HCQ treatment in the last 12 weeks Stop block: stable HCQ treatment for at least the last 12 weeks
5. Ability of subject or/and legal representatives to understand character and individual consequences of clinical trial.
6. Signed and dated informed consent of the subject (if subject has the ability) and the representatives (of underaged children) must be available before start of any specific trial procedures.

(*may be diagnosed in the absence of a lung biopsy by characteristic lung lavage cytology (PAS stain, Fe stain), CT pattern or autoantibodies (gliadin, endomysium; cANCA) and clinical course.)

Exclusion criteria:

Subjects presenting with any of the following criteria will not be included in the trial:

* chILD primarily related to developmental disorders
* chILD primarily related to growth abnormalities reflecting deficient alveolarisation
* chILD related to chronic aspiration
* chILD related to immunodeficiency
* chILD related to abnormalities in lung vessel structure
* chILD related to organ transplantation/organ rejection/GvHD
* chILD related to recurrent infections
* Acute severe infectious exacerbations
* Known hypersensitivity to HCQ, or other ingredients of the tablets (lactose-monohydrate, povidone, maize starch, magnesium stearate, hypromellose, macrogol or titanium dioxide (E 171), silicon dioxide or mannitol), to sucrose-octaacetate or sodium saccharine.
* Proven retinopathy or maculopathy
* Glucose-6-phosphate-dehydrogenase deficiency resulting in favism or hemolytic anemia
* Myasthenia gravis
* Hematopoetic disorders
* Pregnancy and lactation (Women with childbearing potential have to practice a medically accepted contraception during trial and till three months after the end of the treatment with HCQ, and a negative pregnancy test (serum or urine) should be existent on Visit 1, if girls of childbearing age and only if sexual relations are known or probable. It is at the discretion and responsibility of the attending physician to decide, whether a pregnancy test is necessary or not. Reliable contraception are systematic contraceptives (oral, implant, injection). Women that are sterile by surgery can participate in the trial. At the discretion of the investigator, sexual abstinence is also accepted as contraceptive method. Girls after menarche have to receive a counselling about birth control methods in presence of at least one parent, which has to be documented in the patient notes.
* Participation in other clinical trials during the present clinical trial or not beyond the time of 4 half-lives of the medication used, at least one week.
* Hereditary galactose intolerance, lactase deficiency or glucose-galactose- malabsorption
* Renal insufficiency at screening, defined as glomerular filtration rate (GFR)

  * < 40 mL/min/1.73 m2 in patients age 3 to 8 weeks
  * < 60 mL/min/1.73 m2 in patients ≥ 8 weeks of age (KDIGO guideline 2012, K/DOQI guideline 2002)
* Liver disease, gastrointestinal disorder, haematological disorder, epilepsy or other neurological disorder, psoriasis, porphyria at the discretion of the treating physician
* Simultaneous prescription of other potentially nephrotoxic or hepatotoxic medication at the discretion of the treating physician

Ages: 3 Weeks to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Griese, Principal Investigator — Hauner Children´s Hospital, LMU
Locations (9):
- Germany (9):
  - Universitätsklinik für Kinder- und Jugendmedizin Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum der Universität München, Haunersches Kinderspital, München, Bavaria
  - Universitätsklinikum Frankfurt, Pneumologie, Allergologie, Mukoviszidose, Frankfurt am Main, Hesse
  - Justus-Liebig-Universität, Allgemeine Pädiatrie u. Neonatologie, Giessen, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - St. Joseph- und St. Elisabeth Hospital gGmbH, Bochum, North Rhine-Westphalia
  - Uniklinikum Essen, Pädiatrische Pneumologie, Essen, North Rhine-Westphalia
  - Klinik u. Poliklinik für Kinder- u. Jugendmedizin der Universität Leipzig, Leipzig, Saxony
  - Charité Berlin, Klinik für Pädiatrie, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griese M, Kohler M, Witt S, Sebah D, Kappler M, Wetzke M, Schwerk N, Emiralioglu N, Kiper N, Kronfeld K, Ruckes C, Rock H, Anthony G, Seidl E. Prospective evaluation of hydroxychloroquine in pediatric interstitial lung diseases: Study protocol for an investigator-initiated, randomized controlled, parallel-group clinical trial. Trials. 2020 Apr 3;21(1):307. doi: 10.1186/s13063-020-4188-4. PMID 32245508
- [Background] Braun S, Ferner M, Kronfeld K, Griese M. Hydroxychloroquine in children with interstitial (diffuse parenchymal) lung diseases. Pediatr Pulmonol. 2015 Apr;50(4):410-9. doi: 10.1002/ppul.23133. Epub 2014 Dec 9. PMID 25491573
- [Result] Griese M, Kappler M, Stehling F, Schulze J, Baden W, Koerner-Rettberg C, Carlens J, Prenzel F, Nahrlich L, Thalmeier A, Sebah D, Kronfeld K, Rock H, Ruckes C; HCQ-study group; Wetzke M, Seidl E, Schwerk N. Randomized controlled phase 2 trial of hydroxychloroquine in childhood interstitial lung disease. Orphanet J Rare Dis. 2022 Jul 23;17(1):289. doi: 10.1186/s13023-022-02399-2. PMID 35871071

RESULTS

PARTICIPANT FLOW:
Groups:
- Start Placebo, Then HCQ: Placebo for 4 weeks in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg (Group A).
  Followed by Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg. (Group C).
- Start HCQ, Then HCQ: Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg (Group B).
  Followed by HCQ for 4 weeks (Group D)
- Stop HCQ, Then no Medication: Individual dose, usually Hydroxychloroquine Sulfate (HCQ, Quensyl) 6-10 mg/kg bw/d, p.o., one daily dose in the evening; the maximum daily dose is 400 mg. The dose, on which the patient is included into the trial, was continued for 3 months. After therapy of 3 months the medication will be stopped. (Group E) The patient will be followed up for additional 3 months on no medication. (Group G)
- Stop Placebo, Then no Medication: PLACEBO (given according to the individual dose the patient used to take as usually Hydroxychloroquine Sulfate (HCQ, Quensyl) before 6-10 mg/kg bw/d, p.o., one daily dose in the evening; the maximum daily dose is 400 mg. The dose, on which the patient is included into the trial, was continued for 3 months. After therapy of 3 months the PLACEBO will be stopped. (Group F) The patient will be followed up for additional 3 months on no medication. (Group H)
Period: First 4 Wks Start, First 3 Mon Stop
Arm/Group | Start Placebo, Then HCQ | Start HCQ, Then HCQ | Stop HCQ, Then no Medication | Stop Placebo, Then no Medication
Started | 17 | 9 | 4 | 5
Completed | 13 | 7 | 3 | 5
Not Completed | 4 | 2 | 1 | 0
Not completed — Physician Decision | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Second 4 Wks Start, 2nd 3 Mon Stop
Arm/Group | Start Placebo, Then HCQ | Start HCQ, Then HCQ | Stop HCQ, Then no Medication | Stop Placebo, Then no Medication
Started | 13 | 7 | 3 | 5
Completed | 12 | 7 | 3 | 5
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Start Placebo (Group A), Then Continue HCQ (Group C): Placebo for 4 weeks in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg (Group A).
  Followed by Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg. (Group C).
- Start HCQ (Group B), Then Continue HCQ (Group D): Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg (Group B).
  Followed by HCQ for 4 weeks (Group D)
- Stop HCQ (Group E), Then Continued no Medication (Group G): Individual dose, usually Hydroxychloroquine Sulfate (HCQ, Quensyl) 6-10 mg/kg bw/d, p.o., one daily dose in the evening; the maximum daily dose is 400 mg. The dose, on which the patient is included into the trial, was continued for 3 months. After therapy of 3 months the medication will be stopped. (Group E) The patient will be followed up for additional 3 months on no medication. (Group G)
- Stop Placebo (Group F), Then Continued no Medication (Group H): PLACEBO (given according to the individual dose the patient used to take as usually Hydroxychloroquine Sulfate (HCQ, Quensyl) before 6-10 mg/kg bw/d, p.o., one daily dose in the evening; the maximum daily dose is 400 mg. The dose, on which the patient is included into the trial, was continued for 3 months. After therapy of 3 months the PLACEBO will be stopped. (Group F) The patient will be followed up for additional 3 months on no medication. (Group H)
- Total: Total of all reporting groups
Arm/Group | Start Placebo (Group A), Then Continue HCQ (Group C) | Start HCQ (Group B), Then Continue HCQ (Group D) | Stop HCQ (Group E), Then Continued no Medication (Group G) | Stop Placebo (Group F), Then Continued no Medication (Group H) | Total
Number analyzed (Participants) | 17 | 9 | 4 | 5 | 35
Age, Customized [Number; unit: n amount of patients] | 9 | 7.8 | 8.2 | 9.2 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 2 | 3 | 22
  Male | 7 | 2 | 2 | 2 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 16 | 9 | 4 | 5 | 34
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 17 | 9 | 4 | 5 | 35
O2 sat [%] [Number; unit: % 02 saturation] | 92.6 | 93.9 | 93.7 | 94.8 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygenation (Presence or Absence of Response to Treatment) Defined as Change in O2 Saturation >=5%, or Change in Respiratory Rate >=20%, or Change in Respiratory Support Necessary
Description: O2 saturation measured after 5 min at rest and after withdrawal of oxygen if supplied. Change in Oxygenation (presence or absence of response to treatment) defined as change in O2 saturation >=5%, or change in respiratory rate >=20%, or change in respiratory support necessary
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: Group D received HCQ for 4 weeks. These patients had also previously as group B 4 weeks of HCQ, thus an exposure of 8 weeks. This was not deemed comparable to 4 weeks of placebo. Group H received no medication for 3 months. These patients had already withdrawal of HCQ for 3 months as group F, thus no HCQ exposure for 6 months. This was not deemed comparable to 3 months on HCQ. The data of groups D and H were thus not used for the indicated statistical comparisons.
Measure: Count of Participants; unit: Participants
Groups:
- Start Placebo, Then HCQ (Group A): Placebo for 4 weeks in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg.
- Start HCQ, Then HCQ (Group B): Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg (Group B).
- Start Placebo, Then HCQ (Group C): (After 4 weeks of Placebo) now followed by Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg.
- Start HCQ, Then HCQ (Group D): (After 4 weeks of HCQ) now followed by (further) HCQ for 4 weeks
- Stop HCQ, Then no Medication (Group E): Individual dose, usually Hydroxychloroquine Sulfate (HCQ, Quensyl) 6-10 mg/kg bw/d, p.o., one daily dose in the evening; the maximum daily dose is 400 mg. The dose, on which the patient is included into the trial, was continued for 3 months. After therapy of 3 months the medication will be stopped.
- Stop Placebo, Then no Medication (Group F): PLACEBO (given according to the individual dose the patient used to take as usually Hydroxychloroquine Sulfate (HCQ, Quensyl) before 6-10 mg/kg bw/d, p.o., one daily dose in the evening; the maximum daily dose is 400 mg. The dose, on which the patient is included into the trial, was continued for 3 months. After therapy of 3 months the PLACEBO will be stopped.
  The patient will be followed up for additional 3 months on no medication. (Group H)
- Stop HCQ, Then no Medication (Group G): Now the patient was followed for additional 3 months on no medication.
- Stop Placebo, Then no Medication (Group H): Then the patient was followed for additional 3 months on no medication. (Group H)
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 7 | 3 | 5 | 3 | 5
Participants
  Responder | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1
  Non-responder | 13 | 7 | 9 | 7 | 3 | 5 | 2 | 4
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 1, Fisher Exact; No estimated value can be calculated if in any group no responder exists (i.e. no odds exists for independent groups)
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Other — McNemar test for paired samples was not calculated as in any group no responder exists (i.e. no odds exists for independent groups or no discordant pairs could be determined for dependent groups); No estimated OR value can be calculated if in any group no responder exists (i.e. no odds exists for independent groups) and no P values can be calculated as in any group no responder existed (i.e. no odds exists for independent groups or no disconcordant pairs could be determined for dependent groups)
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 1.0, Fisher Exact; No estimated value can be calculated if in any group no responder exists (i.e. no odds exists for independent groups)
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Other — [test comment as in outcome 1, analysis 2]; [other analysis details as in outcome 1, analysis 2]

2. Secondary Outcome: Change in Oxygenation (Presence or Absence of Response to Treatment) Defined as Change in O2 Saturation >=3%, or Change in Respiratory Rate >=20%, or Change in Respiratory Support Necessary
Description: O2 saturation measured after 5 min at rest and after withdrawal of oxygen if supplied. Change in Oxygenation (presence or absence of response to treatment) defined as change in O2 saturation >=3%, or change in respiratory rate >=20%, or change in respiratory support necessary
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Start Placebo, Then HCQ (Group C): Now followed by Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg bw/d, p.o., one daily dose in the evening for 7 days, then reduction to 6.5 mg/kg bw/d for 3 weeks; the maximum daily dose is 400 mg.
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 6 | 12 | 6 | 3 | 5 | 3 | 5
Participants
  Responder | 2 | 1 | 2 | 0 | 0 | 3 | 1 | 1
  Non-responder | 11 | 5 | 10 | 6 | 3 | 2 | 2 | 4
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 1.0, Fisher Exact; Odds Ratio (OR) = 1, 1.1% CI 2-sided [0.079 to 15.16]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 1.0, McNemar; Odds Ratio (OR) = -0.2, 95% CI 2-sided [-0.340 to 0.008]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.196, Fisher Exact; No estimated value can be calculated if in any group no responder exists (i.e. no odds exists for independent groups)
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Other — [test comment as in outcome 1, analysis 2]; [other analysis details as in outcome 1, analysis 2]

3. Secondary Outcome: Change of O2-sat in Room Air (%)
Description: Oxygen saturation in room air at rest
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of O2 Sat
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 6 | 3 | 5 | 3 | 5
percentage of O2 Sat | -0.1 (2.4) | -0.6 (3.3) | 1.8 (3.5) | -1.7 (2.6) | 0.3 (1.2) | -2.4 (2.7) | -3.7 (6.4) | 0.2 (4.8)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.757, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.229, t-test, 2 sided; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.2 to 1.1]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.097, t-test, 2 sided; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.7 to 0.4]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Superiority; p = 0.427, t-test, 2 sided; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.5 to 0.8]

4. Secondary Outcome: Change of Respiratory Rate in Room Air (Breaths/Min)
Description: Respiratory rate in room air at rest measured in breaths per minute
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 5 | 3 | 5 | 3 | 5
breaths/min | 1.2 (5.4) | 0.2 (0.4) | -1.3 (5.6) | 13.8 (33.1) | -2.7 (1.2) | -5.4 (9.4) | 7.3 (5) | 2.5 (7.9)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.543, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.421, t-test, 2 sided; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.553, t-test, 2 sided; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.8 to 1.1]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group H); Test type: Superiority; p = 0.1020, t-test, 2 sided; Mean Difference (Net) = -2.8, 95% CI 2-sided [-5 to -0.5]

5. Secondary Outcome: Change of Quality of Life (chILD Specific)
Description: Quality of life (chILD specific) questionaire. A 5-point response scale was utilized (0 = never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem). Items were reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). Higher scores indicate better HrQoL.
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 2 | 3 | 5 | 3 | 3
score on a scale | 6.9 (9.6) | 0.1 (3.18) | -3.2 (4.8) | -9.1 (3.25) | -5.7 (11.2) | 7.5 (2.3) | 2.3 (3.2) | -2.0 (12.3)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.178, t-test, 2 sided; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.4 to 0.9]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.110, t-test, 2 sided; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.6 to -0.1]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.338, t-test, 2 sided; Mean Difference (Net) = 1.6, 95% CI 2-sided [-0.6 to 3.9]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G) vs Stop Placebo, Then no Medication (Group H); Test type: Superiority; p = 0.3979, t-test, 2 sided; Mean Difference (Net) = -1.0, 95% CI 2-sided [-3 to 1.1]

6. Secondary Outcome: Change of Quality of Life (Total Score)
Description: Quality of life (total score) questionaire. A 5-point response scale was utilized (0 = never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem). Items were reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). Higher scores indicate better HrQoL.
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 3 | 3 | 5 | 3 | 3
score on a scale | 0.4 (6.9) | 0.3 (1.2) | 4.8 (4.3) | 0.4 (7.0) | 9.2 (5.4) | -9.5 (8.8) | -1.7 (2.3) | -5.5 (4.3)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.965, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [-1.6 to 1.6]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.374, t-test, 2 sided; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.4 to 1.9]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.149, t-test, 2 sided; Mean Difference (Net) = -2.6, 95% CI 2-sided [-5.2 to 0.1]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Superiority; p = 0.2963, t-test, 2 sided; Mean Difference (Net) = 2.6, 95% CI 2-sided [0 to 5.3]

7. Secondary Outcome: Change of BMI Percentile
Description: BMI percentile to adapt for age and sex related differences
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 7 | 3 | 5 | 3 | 5
percentile | 7.5 (11.7) | -1.8 (5.1) | -1.6 (8.1) | 22.6 (43.7) | -3.3 (7.9) | 2.2 (11.4) | 13.3 (20.9) | 3.9 (9.2)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.024, t-test, 2 sided; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.9 to 0]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.045, t-test, 2 sided; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.7 to -0.1]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.458, t-test, 2 sided; Mean Difference (Net) = 0.5, 95% CI 2-sided [-0.9 to 2.0]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Superiority; p = 0.4216, t-test, 2 sided; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.8 to 0.7]

8. Secondary Outcome: Change of LDH (U/ml)
Description: Lactate dehydrogenase
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: There was no blood sampled at the visit at the end of group G and H, thus no values available. Group D received HCQ for 4 weeks. These patients had also previously as group B 4 weeks of HCQ, thus an exposure of 8 weeks. This was not deemed comparable to 4 weeks of placebo. This was not deemed comparable to 3 months on HCQ. The data of groups D and H were thus not used for the indicated statistical comparisons.
Measure: Mean (Standard Deviation); unit: Enzyme activity units per ml
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 9 | 5 | 10 | 6 | 2 | 3 | 0 | 0
Enzyme activity units per ml | -28.2 (53.7) | 43.0 (61) | 11.3 (67) | -32.2 (55.3) | 34.5 (0.7) | 9.3 (65.5) |  |
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.063, t-test, 2 sided; Mean Difference (Net) = 1.3, 95% CI 2-sided [0.1 to 2.5]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.410, t-test, 2 sided; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.3 to 1.6]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.574, t-test, 2 sided; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.3 to 1.3]

9. Secondary Outcome: Absolute Change of Forced Vital Capacity (FVC) (% Predicted of the Reference Population)
Description: FVC predicted expressed in % of the normal reference population (Quanjer PH, Brazzale DJ, Boros PW, et al. Implications of adopting the Global Lungs Initiative 2012 all-age reference equations for spirometry. Eur Respir J. 2013;42:1046-54.) The absolute change in FVC % predicited between two measurements is reported.
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of reference population
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 4 | 3 | 5 | 3 | 2
percentage of reference population | 0.0 (3.7) | 2.5 (13) | 10.6 (19.7) | -1.0 (4.2) | 2.3 (7.6) | 0.5 (2.1) | -1.3 (5.1) | 4.5 (4.9)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.730, t-test, 2 sided; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.9 to 1.5]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.170, t-test, 2 sided; Mean Difference (Net) = 0.7, 95% CI 2-sided [-0.3 to 1.8]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.724, t-test, 2 sided; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.1 to 1.5]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Superiority; p = 0.487, t-test, 2 sided; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.2 to 1.1]

10. Secondary Outcome: Absolute Change of Forced Expiratory Volume in One Second (FEV1) (% Predicted of the Reference Population)
Description: FEV1 predicted expressed in % of the normal reference population (Quanjer PH, Brazzale DJ, Boros PW, et al. Implications of adopting the Global Lungs Initiative 2012 all-age reference equations for spirometry. Eur Respir J. 2013;42:1046-54.). The absolute change in FEV1 % predicited between two measurements is reported.
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of reference population
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 4 | 3 | 5 | 3 | 2
percentage of reference population | 0.6 (4.1) | 2.0 (13.1) | 9.0 (18.6) | 0.5 (5.1) | 0.0 (4.4) | -0.5 (0.7) | -1.0 (4.4) | 5.5 (4.9)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.850, t-test, 2 sided; Mean Difference (Net) = 0.2, 95% CI 2-sided [-1 to 1.4]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.258, t-test, 2 sided; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.4 to 1.6]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.862, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.9 to 1.7]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Superiority; p = 0.840, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.8 to 1.4]

11. Secondary Outcome: Absolute Change of Mean Expiratory Flow Between 25 and 75% of Vital Capacity (MEF25-75) (% Predicted of the Reference Population)
Description: MEF25-75 predicted expressed in % of the normal reference population (Quanjer PH, Brazzale DJ, Boros PW, et al. Implications of adopting the Global Lungs Initiative 2012 all-age reference equations for spirometry. Eur Respir J. 2013;42:1046-54.). The absolute change in MEF25-75 % predicited between two measurements is reported.
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of reference population
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 13 | 7 | 12 | 4 | 3 | 5 | 3 | 2
percentage of reference population | 3.0 (13.1) | -14.8 (15.2) | -2.6 (8.6) | 18.5 (17.4) | -8.7 (14.2) | -7.0 (1.4) | -11.3 (7.8) | 15.5 (6.4)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority; p = 0.010, t-test, 2 sided; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.6 to 0]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.533, t-test, 2 sided; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.5 to 0.5]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.858, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.6 to 1.9]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Superiority; p = 0.661, t-test, 2 sided; Mean Difference (Net) = 0.2, 95% CI 2-sided [-1.4 to 1.8]

12. Secondary Outcome: Absolute Change of Six Minute Walking Test (6MWT) Distance (% Predicted of the Reference Population)
Description: 6 Minute walking distance expressed as % of the predicted distance for age and sex. Ulrich et al, Reference values for the 6-minute walk test. BMC Pulm Med. 2013 Aug 5:13:49. doi: 10.1186/1471-2466-13-49. The absolute difference of two measuremnts between two time points is reported.
Time Frame: Start block: A,B after 4 and C,D after 8 weeks; Stop block: E,F after 12 and G,H after 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of reference population
Arm/Group | Start Placebo, Then HCQ (Group A) | Start HCQ, Then HCQ (Group B) | Start Placebo, Then HCQ (Group C) | Start HCQ, Then HCQ (Group D) | Stop HCQ, Then no Medication (Group E) | Stop Placebo, Then no Medication (Group F) | Stop HCQ, Then no Medication (Group G) | Stop Placebo, Then no Medication (Group H)
Number analyzed (Participants) | 4 | 1 | 4 | 1 | 3 | 2 | 3 | 2
percentage of reference population | -0.8 (3.6) | -31.0 (NA) — n.a. because with n=1 you cannot calculate SD | 0.8 (2.1) | 44 (NA) — n.a. because with n=1 you cannot calculate SD | 0.3 (8.5) | -0.5 (2.1) | 8.7 (12.6) | -3.0 (2.8)
Statistical Analysis 1: Comparison: Start Placebo, Then HCQ (Group A) vs Start HCQ, Then HCQ (Group B); Test type: Superiority — Due to missing values no statistical test resulting in a P was calculated; Mean Difference (Net) = -8.4, 95% CI 2-sided [-14 to -2.7]
Statistical Analysis 2: Comparison: Start Placebo, Then HCQ (Group A) vs Start Placebo, Then HCQ (Group C); Test type: Superiority; p = 0.576, t-test, 2 sided; Mean Difference (Net) = 0.5, 95% CI 2-sided [-0.9 to 2]
Statistical Analysis 3: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop Placebo, Then no Medication (Group F); Test type: Superiority; p = 0.884, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.9 to 1.7]
Statistical Analysis 4: Comparison: Stop HCQ, Then no Medication (Group E) vs Stop HCQ, Then no Medication (Group G); Test type: Superiority; p = 0.563, t-test, 2 sided; Mean Difference (Net) = 0.8, 95% CI 2-sided [-2.4 to 0.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected separately according their occurance during Start periods (8 weeks) or Stop periods (6 months).
Description: Adverse events were collected based on the initial assignment in the START or STOP arms. This resulted in the START arm in an allocation of AEs under HCQ to placebo (only group C) and in the STOP arm of placebo events to HCQ (only group G). This mistake was noticed after closure of the data analysis, when entering into Clin.gov. The overall type and frequency of AEs are correct, the frequencies allocated HCQ may be underestimated and those for placebo overestimated. The SAE occurred in group A.
Groups:
- Stop Placebo, Then no Medication: lacebo (given according to the individual dose the patient used to take as usually Hydroxychloroquine Sulfate (HCQ, Quensyl) before 6-10 mg/kg bw/d, p.o., one daily dose in the evening; the maximum daily dose is 400 mg. The dose, on which the patient is included into the trial, was continued for 3 months. After therapy of 3 months the placebo will be stopped. (Group F) The patient will be followed up for additional 3 months on no medication. (Group H)
Arm/Group | Start Placebo, Then HCQ | Start HCQ, Then HCQ | Stop HCQ, Then no Medication | Stop Placebo, Then no Medication
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/7 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 12/13 | 7/7 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Start Placebo, Then HCQ (N=13) | Start HCQ, Then HCQ (N=7) | Stop HCQ, Then no Medication (N=4) | Stop Placebo, Then no Medication (N=5)
Placebogroup Startarm SAE due to infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This occurred in the placebo group in a sick infant on non-invasive respiratory support who had to be intubated due to an intercurrent infection. The SAE resolved completely.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Start Placebo, Then HCQ (N=13) | Start HCQ, Then HCQ (N=7) | Stop HCQ, Then no Medication (N=4) | Stop Placebo, Then no Medication (N=5)
AEs gastrointestinal disorder (Infections and infestations) | 2 (3) | 2 (4) | 2 (2) | 1 (1) — Constipation, stomatitis
AE General disorders (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — pyrexia, hyperthermia, exercise tolerance decreased
Infections (Infections and infestations) | 9 (14) | 3 (4) | 2 (6) | 4 (13) — Sinusitis, otitis, upper and lower respiratory tract infections
AE Blood (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AE psychiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — restlessness
AE Nervouse System (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AE Eye disorders (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Cataract
AE Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) — Arthralgia
AE respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 2 (2) | 1 (1) — cough, pain

LIMITATIONS AND CAVEATS:
Limitations include not reaching the target number of participants. As this was the first randomized controlled trial in fibrosing chILD performed ever, the study was exploratory and there was no formal sample size calculation. Including more patients was prevented by interference with an authority inspection, COVID19 pandemic and the ultra-rare conditions targeted. See for more details Orphanet J Rare Dis. 2022 Jul 23;17(1):289. doi: 10.1186/s13023-022-02399-2. PMID: 35871071.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT02615938/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT02615938/SAP_001.pdf